CLINICAL TRIAL: NCT04311086
Title: Global Clinical Study of Renal Denervation in the Distal Main and First Order Branch Renal Arteries Using the Symplicity Spyral™ Multi-electrode Renal Denervation System (SPYRAL DYSTAL)
Brief Title: SPYRAL DYSTAL Renal Denervation Global Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPYRAL DYSTAL
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Uncontrolled hypertension; Renal denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Renal Denervation (Experimental): Renal angiography and Renal Denervation (Symplicity Spyral™ multi-electrode renal denervation system)
  Interventions: Device: Renal Denervation (Symplicity Spyral™)

INTERVENTIONS:
Device: Renal Denervation (Symplicity Spyral™) — Device: Symplicity Spyral™ multi-electrode renal denervation system. After a renal angiography according to standard procedures, subjects are treated with the renal denervation procedure.
  Other Names: Renal Angiography; Renal Denervation

SUMMARY:
The objective of this single arm interventional study is to determine if renal denervation performed in the distal main and first order branch renal arteries is as effective in reducing blood pressure as the procedural approach used in the SPYRAL HTN-OFF MED clinical study.

ELIGIBILITY:
Inclusion Criteria:

- Individual has office systolic blood pressure (SBP) ≥ 150 mmHg and <180 mmHg and a diastolic blood pressure (DBP) ≥ 90 mmHg after being off medications.

* Individual has 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP ≥ 140 mmHg and < 170 mmHg.
* Individual is willing to discontinue current antihypertensive medications

Exclusion Criteria:

* Individual has estimated glomerular filtration rate (eGFR) of <45.
* Individual has type 1 diabetes mellitus or poorly-controlled type 2 diabetes mellitus.
* Individual has one or more episodes of orthostatic hypotension.
* Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to become pregnant.
* Individual has frequent intermittent or chronic pain that results in treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment.
* Individual has stable or unstable angina within 3 months of enrollment, myocardial infarction within 3 months of enrollment; heart failure, cerebrovascular accident or transient ischemic attack, or atrial fibrillation at any time.
* Individual works night shifts.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David P Lee, MD, Principal Investigator — Stanford University; Andrew Sharp, MD, Principal Investigator — University Hospital of Wales
Locations (8):
- United States (3):
  - Stanford Hospital and Clinics, Stanford, California
  - Piedmont Heart Institute, Atlanta, Georgia
  - Baylor Heart & Vascular Hospital, Dallas, Texas
- Germany (3):
  - Universitaetsklinikum Erlangen, Erlangen
  - Universitaetsklinikum des Saarlandes, Homburg
  - Herzzentrum Leipzig, Leipzig
- Hippokration General Hospital of Athens, Athens, Greece
- University Hospital of Wales, Cardiff, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Comparison of this study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure have been made for several end points and noted in the descriptions.
Period: Overall Study
Arm/Group | Renal Denervation
Started | 128
Completed | 56
Not Completed | 72

BASELINE CHARACTERISTICS:
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 23
  More than one race | 1
  Unknown or Not Reported | 27
Region of Enrollment [Number; unit: participants]
  Greece | 7
  United States | 24
  United Kingdom | 5
  Italy | 6
  Germany | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure (SBP) as Measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: From Baseline (SV2) to 12 months post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 46
mmHg | -16.6 (10.6)

2. Secondary Outcome: Change in Systolic Blood Pressure (SBP) as Measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: From Baseline (SV2) to 3 months post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 53
mmHg | -1.4 (10.0)

3. Secondary Outcome: Change in Office Systolic Blood Pressure (SBP)
Time Frame: From Baseline (SV2) to 3 months post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 55
mmHg | -9.0 (13.9)

4. Secondary Outcome: Change in Office Systolic Blood Pressure (SBP)
Time Frame: From Baseline (SV2) to 12 months post-procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
mmHg | -20.3 (16.3)

5. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) as Measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: From Baseline (SV2) to 3 months post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 53
mmHg | -1.1 (7.5)

6. Secondary Outcome: Change in Diastolic Blood Pressure (DBP) as Measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Time Frame: From Baseline (SV2) to 12 months post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 46
mmHg | -11.2 (8.2)

7. Secondary Outcome: Change in Office Diastolic Blood Pressure (DBP)
Time Frame: From Baseline (SV2) to 3 month post-procedure
Population: Subjects with evaluable data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 55
mmHg | -4.1 (8.5)

8. Secondary Outcome: Change in Office Diastolic Blood Pressure (DBP)
Time Frame: From Baseline (SV2) to 12 months post-procedure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
mmHg | -9.8 (10.8)

9. Secondary Outcome: Incidence of Achieving Target Office Systolic Blood Pressure (SBP)
Description: Target blood pressure defined as <140 mmHg office Systolic Blood Pressure (SBP)
Time Frame: 3 months post-procedure
Population: Subjects with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 55
Participants | 8

10. Secondary Outcome: Incidence of Achieving Target Office Systolic Blood Pressure (SBP)
Description: Target blood pressure defined as <140 mmHg office Systolic Blood Pressure (SBP)
Time Frame: 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants | 27

11. Secondary Outcome: Acute and Chronic Safety by Evaluating Incidence of Major Adverse Events
Description: Incidence of the following events:
  * All-cause mortality
  * End-stage renal disease (ESRD)
  * Significant embolic event resulting in end-organ damage
  * Renal artery perforation requiring intervention
  * Renal artery dissection requiring intervention
  * Vascular complications
  * Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications or the protocol
  * New renal artery stenosis >70%, confirmed by angiography and as determined by the angiographic core lab at 6 months follow up
Time Frame: From Baseline (SV2) to 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants
  All Cause Mortality | 0
  End-stage renal disease (ESRD) | 0
  Significant embolic event resulting in end-organ damage | 2
  Significant Embolic Event, Kidney | 2
  Renal artery perforation requiring intervention | 0
  Renal artery dissection requiring intervention | 0
  Vascular complications | 0
  Hospitalization for hypertensive crisis | 0
  New renal artery stenosis >70% | 0

12. Secondary Outcome: Incidence of Myocardial Infarction
Description: Defined as the concurrent documentation of two of the three elements listed below in the appropriate clinical circumstance:
  1. Chest pain or ischemic equivalent
  2. New pathologic q waves in at least 2 contiguous ECG leads
  3. Cardiac biomarker elevation by any of the definitions below:
  Appropriate cardiac enzyme data (respecting top-down hierarchy):
  1. CK greater than or equal to 2* URL confirmed by:
     * CKMB > l*URL or
     * in the absence of CKMB: Troponin > l*URL or
  2. in the absence of CK:
     * CKMB > 3*URL
     * In the absence of CK and CKMB: Troponin > 3*URL
     * In the absence of CK, CKMB and Troponin, clinical decision based upon clinical scenario
Time Frame: From baseline (SV2) to 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants | 0

13. Secondary Outcome: Incidence of Stroke
Time Frame: From baseline (SV2) to 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants | 0

14. Secondary Outcome: Incidence of Renal Artery Re-intervention
Description: Interventional procedure performed on the renal artery following completion of the renal denervation procedure and removal of the guide catheter.
Time Frame: From baseline (SV2) to 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants | 0

15. Secondary Outcome: Incidence of Major Bleeding According to TIMI Definition
Description: Intracranial hemorrhage; ≥5g/dl decrease in hemoglobin concentration, a ≥15% absolute decrease in hematocrit, or death due to bleeding within seven days of the procedure)
Time Frame: From baseline (SV2) to 12 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 56
Participants | 0

16. Secondary Outcome: Incidence of Increase in Serum Creatinine >50%
Time Frame: From baseline (SV2) to 12 months post-procedure
Population: Subjects with evaluable data
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation
Number analyzed (Participants) | 53
Participants | 0

17. Other Pre Specified Outcome: Reduction in Systolic Blood Pressure (SBP) Over 24 Hours of ABPM as Measured With 24- Ambulatory Blood Pressure Monitor (ABPM) at 3 Months Post-procedure From Baseline
Description: Comparison of systolic blood pressure reduction over 24 hours of ABPM between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: 3 months post-procedure
Population: 53 Subjects from the SPYRAL DYSTAL study and 153 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with 24-hr SBP change as dependent variable. Treatment and baseline 24-hr SBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 206
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 53
  SPYRAL DYSTAL | -1.4 (10.0)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 153
  SPYRAL HTN-OFF MED | -4.5 (10.8)
Statistical Analysis 1: Comparison: Renal Denervation; Comparison to the SPYRAL HTN-OFF MED study (NCT02439749) using a propensity score stratification (sub classification) adjustment; Test type: Other — A propensity score will be estimated for each patient from a multivariable logistic regression model, which is the probability that the patient is in DYSTAL cohort. In this model, the DYSTAL cohort (binary variable) is the outcome variable, and the following covariates will be considered as independent variables for propensity score analysis model: baseline Office and 24-hour ABPM (continuous) SBP and DBP, age (continuous), gender (dichotomous), BMI (continuous), diabetes (dichotomous); p > 0.05, ANCOVA

18. Other Pre Specified Outcome: Reduction in Diastolic Blood Pressure (DBP) Over 24 Hours as Measured With 24-Ambulatory Blood Pressure Monitor (ABPM) at 3 Months Post-procedure From Baseline
Description: Comparison of diastolic blood pressure reduction over 24 hours of ABPM between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: 3 Months post-procedure
Population: 53 Subjects from the SPYRAL DYSTAL study and 153 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with 24-hr DBP change as dependent variable. Treatment and baseline 24-hr DBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 206
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 53
  SPYRAL DYSTAL | -1.1 (7.5)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 153
  SPYRAL HTN-OFF MED | -3.5 (6.7)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p > 0.05, ANCOVA

19. Other Pre Specified Outcome: Office Systolic Blood Pressure (SBP) Reduction
Description: Comparison of Office Systolic Blood Pressure (SBP) reduction between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: From Baseline (SV2) to 3 months post-procedure
Population: 55 Subjects from the SPYRAL DYSTAL study and 170 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with Office SBP change as dependent variable. Treatment and baseline Office SBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 225
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 55
  SPYRAL DYSTAL | -9.0 (13.9)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 170
  SPYRAL HTN-OFF MED | -9.4 (14.8)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p > 0.05, ANCOVA

20. Other Pre Specified Outcome: Office Diastolic Blood Pressure (DBP) Reduction
Description: Comparison of Office Diastolic Blood Pressure (DBP) reduction between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: From Baseline (SV2) to 3 months post-procedure
Population: 55 Subjects from the SPYRAL DYSTAL study and 170 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with Office DBP change as dependent variable. Treatment and baseline Office DBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 225
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 55
  SPYRAL DYSTAL | -4.1 (8.5)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 170
  SPYRAL HTN-OFF MED | -5.0 (8.3)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p > 0.05, ANCOVA

21. Other Pre Specified Outcome: Procedural Characteristics: Procedure Time (Minutes)
Description: Comparison of procedural characteristics: total procedure duration (minutes) between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: Procedure
Population: 56 Subjects from the SPYRAL DYSTAL study and 182 Subjects from the SPYRAL HTN-OFF MED study (NCT02439749).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Renal Denervation
Number analyzed (Participants) | 238
Minutes
  SPYRAL DYSTAL: number analyzed (Participants) | 56
  SPYRAL DYSTAL | 67.3 (20.6)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 182
  SPYRAL HTN-OFF MED | 99.3 (36.2)

22. Other Pre Specified Outcome: Procedural Characteristics: Denervation Time (Minutes)
Description: Comparison of the procedural characteristics: total denervation time between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: Procedure
Population: 56 Subjects from the SPYRAL DYSTAL study and 182 Subjects from the SPYRAL HTN-OFF MED study (NCT02439749).
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Renal Denervation
Number analyzed (Participants) | 238
Minutes
  SPYRAL DYSTAL: number analyzed (Participants) | 56
  SPYRAL DYSTAL | 35.9 (13.8)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 182
  SPYRAL HTN-OFF MED | 59.7 (24.3)

23. Other Pre Specified Outcome: Procedural Characteristics: Amount of Contrast Used (cc)
Description: Comparison of the procedural characteristics: amount of contrast used (cubic centimeter(cc)) between the SPYRAL DYSTAL study and the SPYRAL HTN-OFF MED study (NCT02439749) who, after a renal angiography according to standard procedures, are treated with the renal denervation procedure.
Time Frame: Procedure
Population: 56 Subjects from the SPYRAL DYSTAL study and 178 Subjects from the SPYRAL HTN-OFF MED study (NCT02439749) with evaluable data.
Measure: Mean (Standard Deviation); unit: (cubic centimeter(cc))
Arm/Group | Renal Denervation
Number analyzed (Participants) | 235
(cubic centimeter(cc))
  SPYRAL DYSTAL: number analyzed (Participants) | 56
  SPYRAL DYSTAL | 172.8 (76.6)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 178
  SPYRAL HTN-OFF MED | 207.8 (96.1)

24. Post Hoc Outcome: Reduction in Systolic Blood Pressure (SBP) Over 24 Hours of ABPM as Measured With 24-Ambulatory Blood Pressure Monitor (ABPM) at 12 Months Post-procedure From Baseline
Description: as for outcome 17
Time Frame: 12 months post-procedure
Population: 46 Subjects from the SPYRAL DYSTAL study and 146 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with 24-hr SBP change as dependent variable. Treatment and baseline 24-hr SBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 192
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 46
  SPYRAL DYSTAL | -16.6 (10.6)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 146
  SPYRAL HTN-OFF MED | -14.3 (11.9)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p < 0.05, ANCOVA

25. Post Hoc Outcome: Reduction in Diastolic Blood Pressure (DBP) Over 24 Hours as Measured With 24-Ambulatory Blood Pressure Monitor (ABPM) at 12 Months Post-procedure From Baseline
Description: as for outcome 18
Time Frame: 12 months post-procedure
Population: 46 Subjects from the SPYRAL DYSTAL study and 146 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with 24-hr DBP change as dependent variable. Treatment and baseline 24-hr DBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 192
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 46
  SPYRAL DYSTAL | -11.2 (8.2)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 146
  SPYRAL HTN-OFF MED | -10.2 (8.2)
Statistical Analysis 1: Comparison: Renal Denervation; Test type: Other — [test comment as in outcome 17, analysis 1]; p < 0.05, ANCOVA

26. Post Hoc Outcome: Office Systolic Blood Pressure (SBP) Reduction
Description: as for outcome 19
Time Frame: From Baseline (SV2) to 12 months post-procedure
Population: 56 Subjects from the SPYRAL DYSTAL study and 171 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with Office SBP change as dependent variable. Treatment and baseline Office SBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 227
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 56
  SPYRAL DYSTAL | -20.3 (16.3)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 171
  SPYRAL HTN-OFF MED | -21.3 (14.2)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p > 0.05, ANCOVA

27. Post Hoc Outcome: Office Diastolic Blood Pressure (DBP) Reduction
Description: as for outcome 20
Time Frame: From Baseline (SV2) to 12 months post-procedure
Population: 56 Subjects from the SPYRAL DYSTAL study and 171 Intent-to-Treat Subjects from the SPYRAL HTN-OFF MED study (NCT02439749). Within each of the 5 strata ANCOVA model with Office DBP change as dependent variable. Treatment and baseline Office DBP as independent variables. In subjects with evaluable data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation
Number analyzed (Participants) | 227
mmHg
  SPYRAL DYSTAL: number analyzed (Participants) | 56
  SPYRAL DYSTAL | -9.8 (10.8)
  SPYRAL HTN-OFF MED: number analyzed (Participants) | 171
  SPYRAL HTN-OFF MED | -10.7 (8.8)
Statistical Analysis 1: Comparison: Renal Denervation; [analysis description as in outcome 17, analysis 1]; Test type: Other — [test comment as in outcome 17, analysis 1]; p > 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were monitored/assessed from subject enrollment (consent) through study exit (up to 12 Months Post Procedure) while Adverse Events were monitored/assessed from subject enrollment (consent) through 6-month visits.
Arm/Group | Renal Denervation
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 7/56
Other Adverse Events (participants affected / at risk) | 38/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=56)
Cardiac arrest (Cardiac disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Arthritis infective (Infections and infestations) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Renal artery dissection (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Renal Denervation (N=56)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (2)
Fatigue (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Swelling face (General disorders) | 1 (1)
Immunisation reaction (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 8 (8)
Diverticulitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Muscle contusion (Injury, poisoning and procedural complications) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 8 (8)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site pain (Injury, poisoning and procedural complications) | 1 (1)
Blood aldosterone increased (Investigations) | 1 (1)
Blood cholesterol increased (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 4 (4)
Blood pressure systolic increased (Investigations) | 1 (1)
Blood testosterone decreased (Investigations) | 1 (1)
Carotid pulse abnormal (Investigations) | 1 (1)
Computerised tomogram kidney abnormal (Investigations) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1)
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dizziness postural (Nervous system disorders) | 1 (1)
Head discomfort (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 10 (10)
Migraine (Nervous system disorders) | 2 (2)
Sciatica (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Stress (Psychiatric disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Nocturia (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 2 (2)
Renal artery dissection (Renal and urinary disorders) | 1 (1)
Renal infarct (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 3 (3)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Essential hypertension (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypertensive crisis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04311086/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT04311086/SAP_002.pdf